CLINICAL TRIAL: NCT01828749
Title: Pelvic CT Imaging in Blunt Trauma: Limiting Low Yield Radiation Exposure in Carefully Selected Adult and Pediatric Patients
Brief Title: Pelvic CT Imaging in Blunt Abdominal Trauma
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 02-13-19E
Record Dates: First submitted 2013-03-13; First posted 2013-04-11 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2015-12

CONDITIONS: Blunt Abdominal Trauma
Keywords: blunt abdominal trauma; CT; radiation exposure, pediatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CT abdomen and pelvis: blunt trauma patients without suspected fractures of the pelvis, hip or lumbar spine in two age groups: ages 3-17 years and 18-60 years

SUMMARY:
Abdominopelvic CT (CTap) utilization rose significantly in blunt trauma patients over the last decade. However, the observed increases failed to reduce mortality or missed injury rates. Several investigators have derived (citation) and validated (citation) clinical decision rules that attempt to identify a subset of low risk pediatric and adult patients in whom abdominopelvic CT imaging can be safely eliminated. Thus far these efforts failed to significantly reduce utilization. The investigators propose an alternative and complimentary strategy to decrease radiation by selectively eliminating the pelvic imaging portion of the abdominopelvic CT in low risk patients. In stable, alert patients without clinically evidence of pelvis or hip fractures, abdominal CT imaging alone (diaphragm to iliac crest) identifies clinically significant intra-abdominal injury (cs-IAI) as accurately as routine abdominopelvic imaging (diaphragm to greater trochanter) and results in a clinically important decrease in radiation exposure. The study will investigate this by comparing the accuracy of an imaging protocol using CT abdomen alone versus CT abdomen and pelvis to detect cs-IAI among stable, blunt trauma patients without suspected pelvis or hip fractures in two age groups: ages 3-17 years and 18-60. Patients will undergo CT imaging as deemed clinically indicated by the treating clinician. Among those who have abdominopelvic CT scans, the study will determine the test characteristics of CT abdomen alone versus CT abdomen plus CT pelvis imaging for the identification of cs-IAI. The reference standard will include initial radiology reports, with structured follow up of indeterminate scans, operative reports, and 7-day medical record review.

DETAILED DESCRIPTION:
Abdominopelvic computed tomography (CTap) utilization rose significantly in blunt trauma patients over the last decade but failed to reduce mortality or missed injury rates.

Primary Hypothesis: In stable, alert patients (GCS > 14) without clinically evident fractures of the pelvis, hip or lumbar spine, CT abdomen (CTa) alone (diaphragm to iliac crest) identifies intra-abdominal injury (IAI) with an accuracy that is not inferior to routine CTap (diaphragm to greater trochanter) with a clinically relevant reduction in radiation exposure.

Primary Aim: Compare the accuracy of CTa alone versus CTap to detect IAI in two age groups: ages 3-17 years and 18-60 years. Blunt trauma patients requiring CTap will be enrolled. Data obtained prior to CT imaging include demographics, injury mechanism, exam and pelvic radiograph findings and FAST results from the trauma evaluation. The original CTap will be digitally reformatted to create matched pairs of de-identified CTa and CTap studies. A board certified study radiologist, blinded to the original CT and clinical outcome, will interpret the CTa studies in injured patients. McNemar's chi-square test will be used to evaluate the null hypothesis for injuries in matched pairs assuming no difference for uninjured patients. Te the test characteristics of the CTa versus CTap will be determined. The reference standard will include initial radiology reports, operative reports, and 7-day medical record review. If the upper limit of the 95% confidence interval for the difference in the performance (accuracy) of CTap and CTa alone is less than 3%, the conclusion will be that CTa alone is not inferior to CTap to diagnose IAI. Secondary Aims: The mean effective doses of radiation will be calculated and compared with reductions up to 50% expected. The study will determine if physicians' pretest probability accurately identifies clinically significant pelvis, hip and lumbar spine fractures (CTp indications) in two age groups: ages 3-17 years and 18-60 years. Using a gestalt pretest probability of ≤ 2% as "negative for injury", and a pretest probability > 2% as "positive for injury", the test characteristics of physician estimation will be determined. The test characteristics and interobserver agreement (Cohen's kappa statistic) of exam findings expected to predict fractures of the pelvis, hip and lumbar spine will be reported separately.

ELIGIBILITY:
Inclusion Criteria:

1. 3-60 years of age evaluated for blunt trauma with a GCS of >14
2. Order of CT abdomen and pelvis imaging

Exclusion Criteria:

1. Patients requiring intubation or suspected neurological injury (defined above)
2. Pregnant patients
3. Intoxicated patients
4. Patients with age defined hypotension
5. Exploratory laparotomy or transfusion during the ED evaluation
6. Non-verbal patients
7. Positive FAST exam
8. Patients with abdominal trauma or surgery in the last month
9. Victims of sexual assault or non-accidental trauma (NAT)
10. Patients with known or suspected fractures of the femur or pelvis prior to CT imaging
11. Patients with hip dislocations

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 3-60 years of age evaluated for blunt trauma with a GCS of >14 Order of CT abdomen and pelvis imaging
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Intrabdominal Injury | 7 days
  Accuracy of CT abdomen alone versus CT abdomen and pelvis to detect IAI among stable, blunt trauma patients without suspected fractures of the pelvis, hip or lumbar spine will be compared. The original abdominopelvic CT will be used to create matched pairs of de-identified and digitally reformatted CT abdomen and CT abdomen and pelvis studies. A board certified study radiologist, blinded to the original CT reading and clinical outcome, will interpret the digitally reformatted CT abdomen studies in all injured patients. McNemar's chi-square test will be used to evaluate the null hypothesis for the percentage of correctly identified injuries in the matched pairs assuming no difference for uninjured patients. The sensitivity, specificity and accuracy of the CT abdomen alone versus CT abdomen and pelvis will be determined. The reference standard will include initial radiology reports, with structured follow up of indeterminate scans, operative reports, and 7-day medical record review.

SECONDARY OUTCOMES:
Radiation Exposure | 7 days
  The radiation exposure for imaging protocols of the CT abdomen alone versus CT abdomen and pelvis for study patients in two age groups will be compared: ages 3-17 years and 18-60 years. Using the reported volume CT dose index (CTDI vol), scan length and age specific coefficients for the abdomen/pelvis region of the body, the mean effective radiation doses for CT abdomen alone versus CT abdomen and pelvis will be calculated and compared.
physicians' pretest probability | 7 days
  Determine if physicians' pretest probability accurately identifies clinically significant pelvis, hip and lumbar spine fractures (clinical indications for CT pelvis) in study patients in two age groups: ages 3-17 years and 18-60 years. Using a gestalt pretest probability of ≤ 2% as "negative for injury", and a pretest probability > 2% as "positive for injury", the test characteristics of physician estimation will be determined. The test characteristics and interobserver agreement (Cohen's kappa statistic) of the physical examination findings known to predict fractures of the pelvis, hip and lumbar spine in alert, stable patients for each age group will be reported separately.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Reynolds, MD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States